CLINICAL TRIAL: NCT06876779
Title: Virtual Reality Based Cognitive Behavioral Therapy for Social Anxiety-Driven Depression Among Youths: A Randomized Controlled Trial
Brief Title: Virtual Reality Based Cognitive Behavioral Therapy for Social Anxiety Among Youths in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Shue Yan University (Other)
Responsible Party: Principal Investigator, Wang Yizhou, Assistant Professor, Hong Kong Shue Yan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SATECH
Record Dates: First submitted 2025-02-14; First posted 2025-03-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-01

CONDITIONS: Social Anxiety Disorder (SAD); Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR arm (Experimental): The intervention comprises six sessions of 60 minutes each. There are six VR scenarios such as a café, MTR, school scene, and classroom. The difficulty levels of these scenarios are determined by several factors: (1) the density and proximity of individuals present, as observed in a café or MTR setting, (2) the presence of familiar individuals, such as acquaintances or classmates who may be encountered and greeted in a school environment, and (3) the level of interaction required, such as engaging in a group discussion within a classroom. Participants have the flexibility to choose a different scenario for each session or repeat a previously selected one.
  Interventions: Behavioral: VR intervention
- Treat-as-usual (No Intervention): Participants in the control group will withhold access to the intervention until after the 3-month follow-up assessment. To prevent confounding effects from relevant concomitant care and interventions, participants will be required to refrain from receiving any other treatments or interventions specifically targeting social phobia during the study period.

INTERVENTIONS:
Behavioral: VR intervention — The intervention comprises six sessions of 60 minutes each. There are six VR scenarios such as a café, MTR, school scene, and classroom. The difficulty levels of these scenarios are determined by several factors: (1) the density and proximity of individuals present, as observed in a café or MTR setting, (2) the presence of familiar individuals, such as acquaintances or classmates who may be encountered and greeted in a school environment, and (3) the level of interaction required, such as engaging in a group discussion within a classroom. Participants have the flexibility to choose a different scenario for each session or repeat a previously selected one.
  Arms: VR arm

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a VR-based CBT intervention for social anxiety-driven depression among Hong Kong youth (ages 15-24). Given the limitations of traditional CBT in addressing deep-seated fears, this study explores a more engaging and scalable alternative. Ninety participants with depressive symptoms and social difficulties will undergo six 60-minute VR sessions based on Clark and Wells' cognitive model of social phobia, with assessments at baseline, post-treatment, and three-month follow-up using the Social Phobia Inventory and PHQ-9. The study investigates whether VR intervention reduces social anxiety-driven depression and assesses its cost-effectiveness. Expected outcomes include symptom reduction, sustained benefits at follow-up, and evidence for VR as an innovative, scalable mental health intervention, informing clinical practice, research, and policy in Hong Kong and beyond.

DETAILED DESCRIPTION:
Background: Youth depression in Hong Kong is a growing concern, with a significant number of secondary school and college students exhibiting depressive symptoms. Social anxiety-driven depression, particularly prevalent in this demographic, poses a complex clinical challenge. Current interventions such as cognitive behavioral therapy (CBT), while promising, have limitations in addressing deep-seated fears that hinder engagement in crucial behavioral experiments, and may not fully cater to youth-specific needs.

Method: This study employs a randomized controlled trial design to evaluate the effectiveness of a virtual reality (VR) based CBT intervention in treating social anxiety-driven depression among Hong Kong youths. 90 participants aged 15-24 years, displaying clinical symptoms of depression with self-reported difficulties in social events, will be enrolled. The intervention protocol, grounded in Clark and Wells' cognitive model of social phobia, includes six 60-minute VR sessions simulating various social scenarios. Measurements will be taken at a baseline, post-treatment, and three-month follow-up using tools such as the Social Phobia Inventory and Patient Health Questionnaire-9.

Research Questions: The study primarily investigates whether VR intervention leads to a significant reduction in social anxiety-driven depression post-treatment and follow-ups, as well as the cost analysis of the VR intervention in managing such depression.

Expected Outcomes and Implications: The study anticipates that VR intervention will effectively reduce depression and social anxiety symptoms among participants, with sustained benefits at the three-month follow-up. It is also expected to offer a cost-effective, scalable, and engaging alternative to traditional therapies, addressing a critical gap in youth depression. The findings could have significant implications for academia, practice, providing evidence for the adoption of innovative technology in mental health interventions, and informing future research and policy decisions regarding mental health care for youths in Hong Kong and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. youths aged between 15 and 24 years old; and
2. scoring above 24 on the Social Phobia Inventory.

Exclusion Criteria:

1. unable to attempt a baseline assessment (e.g., due to being unpermitted to leave a psychiatric ward);
2. photosensitive epilepsy;
3. significant visual, auditory, or balance impairment;
4. currently receiving another intensive psychological intervention; and
5. currently holding active suicidal plans

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Social Phobia Inventory (SPIN) | baseline, one-month (post-treatment), and three-month follow-up
  SPIN is a brief self-report tool consisting of 17 items that assess fear, avoidance, and physiological discomfort in social situations. The scale ranges from 0 to 68, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | baseline, one-month (post-treatment), and three-month follow-up
  The Patient Health Questionnaire-9 (PHQ-9) is widely used to screen for the presence and severity of depression, monitor the severity of depression over time, and assist with the diagnosis of depression. The scale ranges from 0 to 27, with higher scores indicating worse outcomes, reflecting greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhou WANG, Assistant Professor, PhD, Principal Investigator — HKSYU

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to ensure participant confidentiality and data security.

REFERENCES:
- [Background] Freeman D, Lister R, Waite F, Galal U, Yu LM, Lambe S, Beckley A, Bold E, Jenner L, Diamond R, Kirkham M, Twivy E, Causier C, Carr L, Saidel S, Day R, Beacco A, Rovira A, Ivins A, Nah R, Slater M, Clark DM, Rosebrock L. Automated virtual reality cognitive therapy versus virtual reality mental relaxation therapy for the treatment of persistent persecutory delusions in patients with psychosis (THRIVE): a parallel-group, single-blind, randomised controlled trial in England with mediation analyses. Lancet Psychiatry. 2023 Nov;10(11):836-847. doi: 10.1016/S2215-0366(23)00257-2. Epub 2023 Sep 21. PMID 37742702
- See also: Related Info — https://www.ugc.edu.hk/eng/rgc/funding_opport/fds/funded%20research/fds2425.html
- Available data/document: Study Protocol — https://www.ugc.edu.hk/eng/rgc/funding_opport/fds/funded%20research/fds2425.html